CLINICAL TRIAL: NCT07063797
Title: Study on the Intervention Effect of Denosumab on High-Risk Patients With Osteoporotic Fractures in Type 2 Diabetes
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2024ZD0532204
Record Dates: First submitted 2025-06-17; First posted 2025-07-14 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-11

CONDITIONS: Type 2 Diabetes; Osteoporosis; Fractures
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Osteoporosis; Fractures, Bone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Denosumab treatment group (Active Comparator): Administer 60 mg of denosumab via subcutaneous injection every six months for a total treatment period of one year.
  Interventions: Drug: Denosumab treatment in type 2 diabetes mellitus (T2DM) with osteoporosis patients
- Denosumab combined with eldecalcitol treatment group (Experimental): Denosumab 60 mg subcutaneous injection, once every six months, combined with eldecalcitol 0.75 μg once daily, for one year of treatment.
  Interventions: Drug: Denosumab combined with eldecalcitol treatment in type 2 diabetes mellitus (T2DM) with osteoporosis patients

INTERVENTIONS:
Drug: Denosumab treatment in type 2 diabetes mellitus (T2DM) with osteoporosis patients — 1. Antihyperglycemic drug therapy: Follow the Chinese Diabetes Treatment Guidelines and clinical practice standards. Adjust the antihyperglycemic regimen based on blood glucose levels, with a target HbA1c of below 7.5%.
  2. Denosumab treatment: Administer 60 mg of denosumab via subcutaneous injection every six months for a total treatment period of one year.
  Arms: Denosumab treatment group
Drug: Denosumab combined with eldecalcitol treatment in type 2 diabetes mellitus (T2DM) with osteoporosis patients — 1. Antihyperglycemic drug therapy: Follow the Chinese Diabetes Treatment Guidelines and clinical practice standards. Adjust the antihyperglycemic regimen based on blood glucose levels, with a target HbA1c of below 7.5%.
  2. Denosumab injection (Mai Lishu), 60 mg subcutaneous injection, once every six months, combined with eldecalcitol soft capsules (Gai Sheng Yuan), 0.75 μg/capsule, take one capsule orally once daily, for one year of treatment.
  Arms: Denosumab combined with eldecalcitol treatment group

SUMMARY:
This study will conduct a randomized controlled trial targeting patients with type 2 diabetes and a high risk of fractures. The aim is to evaluate the intervention effect of denosumab combined with edilossobulin on patients with a high risk of osteoporotic fractures due to type 2 diabetes, as well as its impact on bone density, bone turnover indicators, the risk of new fractures, and the risk of hypocalcemia. This will provide scientific evidence for clinical diagnosis and treatment, and offer important clinical research evidence for formulating national health policies.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of type 2 diabetes (based on the "China Guidelines for the Prevention and Treatment of Diabetes (2024 Edition)").
2. Males aged ≥50 years; females aged ≥45 years and postmenopausal for more than 2 years.
3. Duration of diabetes >10 years; or presence of at least one of the following conditions: ①diabetic retinopathy; ②urine albumin-to-creatinine ratio (UACR)≥ 30 mg/g; ③estimated glomerular filtration rate (eGFR)<60 mL/min/1.73 m²; ④coronary atherosclerotic heart disease; ⑤ischemic stroke; ⑥transient ischemic attack; ⑦ atherosclerosis of the carotid, cerebral, or lower-extremity arteries with ≥50% luminal stenosis.
4. Glycated hemoglobin (HbA1c) ≤ 8.0 % measured within 1 month
5. History of hip or vertebral fragility fractures; or history of fragility fractures at other sites (excluding the skull, feet, and hands) with a T-score of <-1.0 at the femoral neck, total hip, or any L1-L4 site; or a T-score of <-2.0 at the femoral neck, total hip, or any L1-L4 site.
6. In the BMD measurement at lumbar vertebrae L1-L4, at least two or more vertebral bodies must meet the evaluable criteria.
7. Signed informed consent form, willing to participate in the study

Exclusion Criteria:

1. Diseases that cause secondary osteoporosis: a. Various metabolic bone diseases, such as osteomalacia, primary hyperparathyroidism, osteogenesis imperfecta, Paget's disease, etc.; b. Cushing's syndrome; c. Hyperprolactinemia; d. Others;
2. Malignant tumors within the past 5 years, except for those expected to be cured after treatment (e.g., completely resected in situ basal cell or squamous cell carcinoma of the skin, cervical cancer, or ductal carcinoma of the breast);
3. Received intravenous bisphosphonate treatment within the past 2 years or oral bisphosphonate treatment within the past 1 year;
4. History or current diagnosis of osteomyelitis or osteonecrosis of the jaw; unhealed dental or oral surgical wounds; acute dental or jaw conditions requiring oral surgery; planned to undergo invasive dental surgery during the study period;
5. Received denosumab, teriparatide, or romosozumab treatment within the past 6 months;
6. Continuous use of calcitonin for more than 3 months within the past year;
7. Use of glucocorticoids (equivalent to>5 mg/day prednisone) for more than 10 days within the past 6 weeks;
8. 25-hydroxyvitamin D<10ng/mL;
9. Active infections requiring systemic treatment;
10. Uncontrolled comorbidities, including New York Heart Association (NYHA) functional class III or above heart failure, severe arrhythmias, severe hepatic insufficiency (alanine aminotransferase or aspartate aminotransferase>3 times the upper limit of normal), severe renal insufficiency (eGFR<30 ml/min/1.73 m²);
11. Hypocalcemia, hypercalcemia, or hypercalciuria (Note: hypercalciuria is defined as a urinary calcium/creatinine ratio > 0.5 mg/mg, or 24-hour urinary calcium > 7.5 mmol).;
12. Allergy to the study drug;
13. Currently participating in other clinical trials of drugs;
14. Subjects deemed unsuitable for enrollment in this study by the investigator.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 358 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
change rate of lumbar bone density | 12 months of treatment
  DXA measurement

SECONDARY OUTCOMES:
Incidence of osteoporotic fractures | 12 months of treatment
  X ray imaging measurement
Change rate of bone density in the femoral neck and total hip | 12 months of treatment
  DXA measurement
Change rate of serum levels of β-CTX | 6 months of treatment
  electrochemiluminescence measurment
Change rate of serum levels of β-CTX | 12 months of treatment
  electrochemiluminescence measurment
Change rate of serum levels of PINP | 6 months of treatment
  electrochemiluminescence measurment
Change rate of serum levels of PINP | 12 months of treatment
  electrochemiluminescence measurment

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Peking Union Medical College Hospital, Beijing, Dongcheng
  - Huai'an First People's Hospital, Huai'an
  - Jiangxi Provincial People's Hospital, Jiangxi
  - Kunshan Hospital of Traditional Chinese Medicine, Kunshan

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2025-12-05): https://cdn.clinicaltrials.gov/large-docs/97/NCT07063797/Prot_002.pdf
  • Informed Consent Form (2025-12-05): https://cdn.clinicaltrials.gov/large-docs/97/NCT07063797/ICF_003.pdf